CLINICAL TRIAL: NCT01079117
Title: Randomised, Controlled Clinical Study Regarding the Feasibility of Converting Opiate Dependents From Methadone Substitutes to Slow Release Morphine Sulphate (Sevre-Long™)
Brief Title: Morphine Slow-release Capsules in Substitution Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SUB9001; 2008-002185-60 (EudraCT Number)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Opiate Dependent
Keywords: Opiate; Methadone; Slow Release Oral Morphine (SORM); Sevre-Long™
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevre-Long™ (Active Comparator): slow release oral morphine
  Interventions: Drug: Sevre-Long™; Drug: Slow release oral morphine
- Methadone (Active Comparator): Methodone
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Sevre-Long™ — The subjects will be randomised to either 10 weeks of treatment with methadone or SROM. After an adjustment phase of one week they first will be medicated for 10 weeks with the treatment to which they have been randomised. The cross-over, in which all subjects change to their opposite treatment, will serve for an additional adjustment phase of one week. After the second and new adjustment phase they are treated for 10 weeks with the newly adjusted medication. After the end of week 22 all participants continue with or switch back to SROM for another 6 month (week 23 to 47).
  Arms: Sevre-Long™
Drug: Slow release oral morphine
  Arms: Sevre-Long™
Drug: Methadone
  Arms: Methadone

SUMMARY:
To compare the effectiveness of slow release oral morphine treatment in patients that previously have been treated with methadone

DETAILED DESCRIPTION:
The objective of this study is to compare the effectiveness of slow-release oral morphine (SROM) treatment in patients that previously have been treated with methadone. Efficacy is assessed by the frequency of by-consumption of illicit substances. The primary efficacy endpoint in this study is the proportion of positive urine tests for by-consumption of target substances per subject. Target substances are defined as all opioids except the study drug.

The proportions are compared between substitution with methadone and SROM treatment in a crossover design.

The secondary endpoints are:

1. The effects of SROM on retention rate.
2. By-consumption of other drugs (cocaine, alcohol, cannabis, benzodiazepines).
3. Occurring psychopathological and somatic symptoms.
4. Effect of treatment on the ECG (QTc prolongation).
5. Group characterisation of patients that is keen to change the medication.
6. The change in dosage of treatment over time.
7. Self-assessed craving for Opioids.
8. Self-assessed satisfaction with treatment.
9. Nature, frequency and severity of occurring adverse events in the two treatment groups.
10. Assessment of safety parameters.

Study Design (Methodology):

This is a multicentre, multinational phase III study. It is conducted using a randomised, open label cross-over design. The subjects will be randomised to either 10 weeks of treatment with methadone or SROM. After an adjustment phase of one week they first will be medicated for 10 weeks with the treatment to which SUB9001 - Integrated Study Protocol 9/58 June 13, 2009 they have been randomised. The cross-over, in which all subjects change to their opposite treatment, will serve for an additional adjustment phase of one week. After the second and new adjustment phase they are treated for 10 weeks with the newly adjusted medication. After the end of week 22 all participants continue with or switch back to SROM for another 6 month (week 23 to 47).

ELIGIBILITY:
Inclusion criteria:

* Minimum age: 18 years
* Fixed abode
* At least 26 weeks of treatment (up to date) receiving a minimum dose of 50 mg methadone or

  ≥ 25 mg/day levomethadone at inclusion. Patients on levomethadone must be informed and agree to be switched to methadone
* Mature and capable of acting responsibly, in possession of all mental faculties
* Female subjects must have a negative urine pregnancy test recorded prior to the first dose of study medication and regular negative urine pregnancy tests every 4 weeks. SUB9001 - Integrated Study Protocol 10/58 June 13, 2009
* Hormonal contraception (oral, transdermal, vaginal, intrauterine or subcutaneous) by women of child-bearing age
* No intention of reducing the substitute medication during the trial
* Acceptance of the trials rules and regulations
* Acceptance to participate in the study.

Exclusion criteria:

* (Desired) pregnancy during the trial
* Breastfeeding women
* Grave or acute somatic illnesses (e.g. cardio-vascular, serious kidney or liver affection (ALAT or ASAT > 5x augmented)) or other somatic disorder
* If suffering from severe unstable mental health problems
* If MAO-Inhibitors or are being taken
* Intracranial injury
* Intracranial hypertension
* History of epilepsy
* Severe chronic obstructive lung disease
* Chronic respiratory failure
* Known hypersensitivity to morphine or methadone
* Pancreatitis
* Paralytic ileus
* Baseline QTc interval greater than 450 msec
* Long QT Syndrome
* Patients who have participated in another clinical research study involving a new chemical entity within 3 months of study entry
* Patients with pending imprisonment at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2006-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Proportion of positive urine tests for by-consumption of target substances per subject | each week during the 22 week cross-over phase
  The primary efficacy endpoint in this study is the proportion of positive urine tests for by-consumption of target substances per subject.
  Target substances are defined as all opioids except the study drug. The proportions are compared between substitution with methadone and SROM treatment in a crossover design.

SECONDARY OUTCOMES:
Secondary Outcome Measures | throughout the 22 week cross over period
  The effects of SROM on retention rate
By-consumption of other drugs (cocaine, alcohol, cannabis, benzodiazepines) | throughout the 22 week cross over period
Occurring psychopathological and somatic symptoms. | througout the 22 week cross over period
Effect of treatment on the ECG (QTc prolongation) | throughout the 22 week cross over phase
Group characterisation of patients that is keen to change the medication | throughout the 22 week cross over period
The change in dosage of treatment over time | throughout the 22 week cross over period
Self-assessed craving for Opioids | throughout the 22 week cross over period
Self-assessed satisfaction with treatment. | throughout the 22 week cross over period
Nature, frequency and severity of occurring adverse events in the two treatment groups | throughout the 22 week cross over period
Assessment of safety parameters | throughout the 22 week cross over period

CONTACTS AND LOCATIONS:
Locations (1):
- Zurich, Switzerland

REFERENCES:
- [Result] Beck T, Haasen C, Verthein U, Walcher S, Schuler C, Backmund M, Ruckes C, Reimer J. Maintenance treatment for opioid dependence with slow-release oral morphine: a randomized cross-over, non-inferiority study versus methadone. Addiction. 2014 Apr;109(4):617-26. doi: 10.1111/add.12440. Epub 2014 Jan 19. PMID 24304412
- [Derived] Falcato L, Beck T, Reimer J, Verthein U. Self-reported cravings for heroin and cocaine during maintenance treatment with slow-release oral morphine compared with methadone: a randomized, crossover clinical trial. J Clin Psychopharmacol. 2015 Apr;35(2):150-7. doi: 10.1097/JCP.0000000000000288. PMID 25679130
- [Derived] Hammig R, Kohler W, Bonorden-Kleij K, Weber B, Lebentrau K, Berthel T, Babic-Hohnjec L, Vollmert C, Hopner D, Gholami N, Verthein U, Haasen C, Reimer J, Ruckes C. Safety and tolerability of slow-release oral morphine versus methadone in the treatment of opioid dependence. J Subst Abuse Treat. 2014 Oct;47(4):275-81. doi: 10.1016/j.jsat.2014.05.012. Epub 2014 Jun 10. PMID 25064422
- See also: Published study results — http://www.ncbi.nlm.nih.gov/pubmed/24304412